CLINICAL TRIAL: NCT06037187
Title: Coagulopathy of Immunodermatologic Diseases The Molecular, Prognostic, and Therapeutic Implications of Crosstalk Between Coagulation, Fibrinolysis, and Inflammation in Immune-Mediated Skin Diseases
Brief Title: Coagulopathy of Immunodermatologic Diseases
Status: Recruiting | Type: Observational
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Other Study IDs: 0016-23-EP
Record Dates: First submitted 2023-08-29; First posted 2023-09-14 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Autoimmune Bullous Dermatosis
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Immune-mediated condition: Participants with an immune-mediated condition
  Interventions: Diagnostic Test: Blood Draw
- Without immune-mediated dermatologic condition: Participants without an immune-mediated dermatologic condition
  Interventions: Diagnostic Test: Blood Draw

INTERVENTIONS:
Diagnostic Test: Blood Draw — Standard coagulation assays (aPTT, INR, ACT), viscoelastic coagulation profiles (rotational thromboelastometry (ROTEM)/thromboelastography (TEG), tPA-challenged ROTEM/TEG), and molecular profiling

SUMMARY:
This study will examine the coagulation and fibrinolysis profiles of those with autoimmune skin diseases. Blood samples will be collected from participants with active/poorly controlled immune-mediated skin diseases and mild/latent/well-controlled immune-mediated skin diseases. A one-time sample from 15 general dermatology outpatients who do not have a known or suspected diagnosis of bullous diseases, immune-mediated dermatologic condition, or cutaneous malignancy will also be collected to serve as control. Blood samples from both participant populations will be analyzed for coagulation and inflammatory markers and compared. The results of this study may help inform future studies on the utility of analyzing coagulation and fibrinolysis profiles of patients with autoimmune skin diseases.

DETAILED DESCRIPTION:
The purpose of this study is to examine the coagulation and fibrinolysis profiles of those with autoimmune skin diseases. This will be accomplished by collecting blood samples from participants with both active/poorly controlled immune-mediated skin diseases and mild/latent/well-controlled immune-mediated skin diseases. A one-time sample will be collected from 15 general dermatology outpatients who do not have a known or suspected diagnosis of bullous diseases, immune-mediated dermatologic condition, or cutaneous malignancy to serve as the control population. Blood samples from both participant populations will be analyzed for coagulation and inflammatory markers and compared. The results of this study may help inform future studies on the utility of analyzing coagulation and fibrinolysis profiles of patients with autoimmune skin diseases.

ELIGIBILITY:
Inclusion Criteria:

1. For the study group: diagnosis of immune-mediated skin disease including but not limited to bullous pemphigoid, pemphigus vulgaris, mucous membrane pemphigoid, cutaneous lupus erythematosus, dermatomyositis
2. For control group: no diagnosis of immune-mediated skin
3. For study group: receiving care from one or more of the Principal or Secondary Investigators

Exclusion Criteria:

1. Unfit to provide consent
2. P2Y12 inhibitor use in the past 4 weeks
3. History of internal malignancy prior to enrolling in the study or suspected internal/systemic malignancy during time of the study (i.e. will not exclude pre-malignant or local, early stage cutaneous malignancies)
4. Major surgery within 4 weeks of the study or trauma (e.g., accident-causing bone fracture) within 4 weeks of the study
5. Other autoimmune diseases not in remission defined as flare in the last 12 weeks
6. If patient is unable to provide detailed history and if we do not have sufficient history on record.
7. Less than 19 years of age

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients seen at University of Nebraska Medical Center diagnosed with autoimmune bullous disease and patients without a autoimmune bullous disease.
Sampling Method: Non-Probability Sample
Enrollment: 39 (Estimated)
Dates: Start 2023-05-09 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Thromboelastography | 2 years
  Thromboelastography is a viscoelastic hemostatic assay that measures the global viscoelastic properties of whole blood clot formation under low shear stress.
tPA-challenged Thromboelastography | 2 years
  Tests patients blood resistance to tPA-mediated clot lysis.
Activated partial thromboplastin time | 2 years
  Activated partial thromboplastin time measures the length of time (in seconds) that it takes for clotting to occur when specific reagents are added to plasma.
International normalized ratio | 2 years
  International Normalized Ratio is a measure of how long it takes your blood to clot.

CONTACTS AND LOCATIONS:
Overall Officials: Erin X Barrett, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No